CLINICAL TRIAL: NCT02951429
Title: A Phase IIb, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Sildenafil Added to Pirfenidone in Patients With Advanced Idiopathic Pulmonary Fibrosis and Intermediate or High Probability of Group 3 Pulmonary Hypertension
Brief Title: Efficacy, Safety, and Tolerability Study of Pirfenidone in Combination With Sildenafil in Participants With Advanced Idiopathic Pulmonary Fibrosis (IPF) and Intermediate or High Probability of Group 3 Pulmonary Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MA29957; 2015-005131-40 (EudraCT Number)
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Results first posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pirfenidone; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Pirfenidone + Placebo (Placebo Comparator): Participants will receive pirfenidone along with placebo matched to sildenafil, orally, three times a day (TID) for 52 weeks.
  Interventions: Drug: Pirfenidone; Drug: Placebo
- Pirfenidone + Sildenafil (Experimental): Participants will receive pirfenidone along with sildenafil, orally, TID for 52 weeks.
  Interventions: Drug: Pirfenidone; Drug: Sildenafil

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone will be given in the range of 1602 to 2403 milligram per day (mg/day), as 3 divided doses.
  Other Names: Esbriet, RO0220912
Drug: Placebo — Placebo matched with sildenafil.
  Arms: Pirfenidone + Placebo
Drug: Sildenafil — Sildenafil will be given as 20 mg, TID.
  Other Names: RO0280296
  Arms: Pirfenidone + Sildenafil

SUMMARY:
This Phase IIb, randomized, placebo-controlled, multicenter, international study will evaluate the efficacy, safety, and tolerability of sildenafil or placebo added to pirfenidone (Esbriet) treatment in participants with advanced IPF and intermediate or high probability of Group 3 pulmonary hypertension (PH) who are on a stable dose of pirfenidone with demonstrated tolerability. Participants will be randomized to receive 1 year of treatment with either oral sildenafil or matching placebo while continuing to take pirfenidone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPF for at least 3 months prior to Screening
* Confirmation of IPF diagnosis by the investigator in accordance with the 2011 international consensus guidelines at screening
* Advanced IPF (defined as a measurable carbon monoxide diffusing capacity [DLCO] less than or equal to (<=)40% of predicted value at Screening) and intermediate or high probability of group 3 pulmonary hypertension (PH)
* Participants receiving pirfenidone for at least 12 weeks, at a dose in the range of 1602 to 2403 mg/day for at least 4 weeks prior to Screening and must not have experienced either a new or ongoing adverse event of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (version 4.03) Grade 2 or higher and considered by the investigator to be related to pirfenidone, or an interruption of pirfenidone treatment of greater than (>)7 days for any reason
* WHO Functional Class II or III at Screening
* 6MWD of 100 to 450 meters at screening
* Women of childbearing potential and for men who are not surgically sterile agreement to remain abstinent or use of contraceptive measures

Exclusion Criteria:

* History of any of the following types of PH: Group 1 (PAH); Group 1 (pulmonary veno-occlusive disease and/or pulmonary capillary hemangiomatosis); Group 2 (left-heart disease); Group 3 (due to conditions other than interstitial lung disease, including chronic obstructive pulmonary disease [COPD], sleep-disordered breathing, alveolar hypoventilation, high altitude, or developmental abnormalities); Group 4 (chronic thromboembolic pulmonary hypertension); Group 5 (other disorders)
* History of clinically significant cardiac disease
* History of coexistent and clinically significant COPD, bronchiectasis, asthma, inadequately treated sleep-disordered breathing, or any clinically significant pulmonary diseases or disorders other than IPF or PH secondary to IPF
* History of use of drugs and toxins known to cause PAH, including aminorex, fenfluramine, dexenfluramine, and amphetamines
* FEV1/FVC ratio less than (<) 0.70 post bronchodilator; SpO2 saturation at rest <92% with >= 6 liters (L) of supplemental oxygen at Screening
* Extent of emphysema greater than the extent of fibrotic changes (honeycombing and reticular changes) on any previous high-resolution computed tomography (HRCT) scan, in the opinion of the Investigator
* Smoked tobacco within 3 months prior to screening or is unwilling to avoid tobacco products (cigarettes, pipe, cigars) throughout the study
* Illicit drug or significant alcohol abuse
* Electrocardiogram (ECG) with a heart-rate corrected QT interval (corrected using Fridericia's formula [QTcF]) >=500 milliseconds (ms) at screening, or a family or personal history of long QT syndrome
* Exclusion criteria based on pirfenidone reference safety information: 1. participants with a history of angioedema due to pirfenidone; 2. concomitant use of fluvoxamine
* Exclusion criteria based on sildenafil reference safety information: 1. co-administration with nitric oxide donors or organic nitrates, phosphodiesterase-5 (PDE5) inhibitors, guanylate cyclase stimulators, and most potent of the Cytochrome P450 3A4 (CYP3A4) inhibitors; 2. loss of vision in one eye because of non-arteritic anterior ischemic optic neuropathy (NAION); 3. use of an alpha-blocker; 4. participants with bleeding disorders or active peptic ulceration; 5. known hereditary degenerative retinal disorders such as retinitis pigmentosa; 6. galactose intolerance

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2016-12-31 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2020-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (56):
- Belgium (6):
  - ULB Hôpital Erasme, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Antwerpen, Edegem
  - UZ Leuven Gasthuisberg, Leuven
  - CHU Sart-Tilman, Liège
  - CHU UCL Mont-Godinne, Mont-godinne
- Canada (3):
  - Hotel Dieu Hospital, Kingston, Ontario
  - CHUM Hôpital Notre-Dame, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec (Hôpital Laval), Ste. Foy, Quebec
- Thomayerova nemocnice; Pneumologicka klinika 1.LF UK TN, Praha 4 - Krc, Czechia
- Egypt (3):
  - Clinical Research Center (CRC), Faculty of Medicine, Alexandria University, Alexandria
  - Kasr El-Aini-Chest Unit; Department 3-Chest Unit, Cairo
  - Ain Shams University Hospital-Chest unit; Chest unit, Cairo
- Germany (8):
  - Fachkrankenhaus Coswig GmbH Zentrum f.Pneumologie Beatmungsmedizin Thorax-u.Gefäßchirurgie, Coswig
  - Klinik Donaustauf Zentrum für Pneumologie, Donaustauf
  - Ruhrlandklinik Lungenzentrum der UNI Essen Abt.Pneumologie-Allergologie, Essen
  - Klinikum Fulda gAG; Universitätsmedizin Marburg, Campus Fulda, Fulda
  - Universitätsklinikum Standort Gießen Medizinische Klinik II u. Poliklinik Innere Med./Pneumologie, Giessen
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Fachklinik für Lungenerkrankungen, Immenhausen
  - Klinikum der Universität München; Campus Großhadern; Med. Klinik und Poliklinik V, München
- Greece (3):
  - Sotiria Hospital for Diseases of the Chest, Academic Department of Pneumonology, Athens
  - University General Hospital of Athens "Attikon", B' University Pulmonary Clinic, Chaïdári
  - University General Hospital of Heraklio, Pulmonary Clinic, Heraklio
- Hungary (2):
  - Semmelweis Egyetem X; Pulmonologiai Klinika, Budapest
  - Orszagos Koranyi TBC es Pulmonologiai Intezet, Budapest
- Israel (7):
  - Soroka; Pulmonary Clinic, Beersheba
  - Carmel Medical Center; Pulmonary Institute, Haifa
  - Shaare Zedek Medical Center; Pulmonary Inst., Jerusalem
  - Hadassah Medical Center; Pulmonary Institute, Jerusalem
  - Meir Medical Center; Pulmonary Dept, Kfar Saba
  - Beilinson Medical Center; Pulmonary Inst., Petah Tikva
  - Kaplan Medical Center, Rehovot
- Italy (8):
  - A.O.U. Ospedali Riuniti Di Foggia-Ospedale D'avanzo; Malattie Dell'apparato Respiratorio IV, Foggia, Apulia
  - Ospedale Morgagni-Pierantoni; U.O. Pneumologia, Forlì, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena; DIP. Malattie Dell'apparato Respiratorio, Modena, Emilia-Romagna
  - Ospedale San Giuseppe; U.O. di Pneumologia, Milan, Lombardy
  - ASST DI MONZA; U O Clinica Pneumologica, Monza, Lombardy
  - A.O.U. Policlinico Vittorio Emanuele; Centro per la cura delle Malattie Rare del Polmone, Catania, Sicily
  - A.O. Univ. Senese Policlinico S. Maria alle Scotte; UOC Malattie Resepiratorie e Trapianto Polmonare, Siena, Tuscany
  - Azienda Ospedaliera di Padova; Dip. Scienze Cardiologiche Toraciche Vascolari-UOC Pneumologia, Padua, Veneto
- Netherlands (2):
  - Vu Medisch Centrum; Afdeling Longziekten, Amsterdam
  - Erasmus MC, Rotterdam
- South Africa (3):
  - University of Cape Town Lung Institute; Lung Clinical Research, Cape Town
  - Milpark Hospital, Parktown West
  - University of Stellenbosch; Respiratory Research, Parow
- Spain (5):
  - Hospital Universitari de Bellvitge ; Servicio de Neumologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla; Servicio de neumologia, Santander, Cantabria
  - Hospital Universitario Puerta de Hierro Majadahonda; Servicio de Neumología, Majadahonda, Madrid
  - Hospital Clinic I provincial; Servicio de Neumologia, Barcelona
  - Hospital Universitario la Fe; Servicio de Neumologia, Valencia
- Turkey (Türkiye) (5):
  - Ankara Uni Faculty of Medicine; Chest Diseases, Ankara
  - Uludag University; Pulmonology and Allergy Department, Bursa
  - Yedikule Gogus Hastaliklari ve Gogus Cerrahisi EAH;Gogus Hastaliklari, Istanbul
  - Istanbul Universitesi Capa Tıp Fakültesi; Gogus Hastalıkları Anabilim dalı, Istanbul
  - Ege Universitesi Tıp Fakültesi; Gögüs Hastalıkları Bilim Dalı, Izmir

REFERENCES:
- [Derived] Behr J, Nathan SD, Costabel U, Albera C, Wuyts WA, Glassberg MK, Haller H Jr, Alvaro G, Gilberg F, Samara K, Lancaster L. Efficacy and Safety of Pirfenidone in Advanced Versus Non-Advanced Idiopathic Pulmonary Fibrosis: Post-Hoc Analysis of Six Clinical Studies. Adv Ther. 2023 Sep;40(9):3937-3955. doi: 10.1007/s12325-023-02565-3. Epub 2023 Jun 30. PMID 37391667
- [Derived] Behr J, Nathan SD, Wuyts WA, Mogulkoc Bishop N, Bouros DE, Antoniou K, Guiot J, Kramer MR, Kirchgaessler KU, Bengus M, Gilberg F, Perjesi A, Harari S, Wells AU. Efficacy and safety of sildenafil added to pirfenidone in patients with advanced idiopathic pulmonary fibrosis and risk of pulmonary hypertension: a double-blind, randomised, placebo-controlled, phase 2b trial. Lancet Respir Med. 2021 Jan;9(1):85-95. doi: 10.1016/S2213-2600(20)30356-8. Epub 2020 Aug 18. PMID 32822614

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Written informed consent for participation in the study was obtained before performing any study-specific screening tests or evaluations.
Groups:
- Pirfenidone+Sildenafil: Participants received pirfenidone along with sildenafil, orally, three times a day for 52 weeks.
- Pirfenidone+Placebo: Participants received pirfenidone along with placebo matched to sildenafil, orally, three times a day for 52 weeks.
Period: Overall Study
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Started | 88 | 89
Completed | 16 | 6
Not Completed | 72 | 83
Not completed — Adverse Event | 3 | 7
Not completed — Death | 28 | 36
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lung Transplantation | 9 | 6
Not completed — Other | 1 | 3
Not completed — Progressive Disease | 1 | 1
Not completed — Withdrawal by Subject | 7 | 11
Not completed — Participant ongoing in the study | 23 | 17

BASELINE CHARACTERISTICS:
Population: ITT Population -
Groups:
- Total: Total of all reporting groups
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo | Total
Number analyzed (Participants) | 88 | 89 | 177
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.2 (7.7) | 68.9 (7.1) | 68.6 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 43
  Male | 69 | 65 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 78 | 79 | 157
  Unknown or Not Reported | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  White | 85 | 88 | 173
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Progression, as Determined by Relevant Decline in 6 Minute Walk Distance (6MWD) of At Least (>=) 15 Percent (%) From Baseline, Respiratory-Related Non-Elective Hospitalization, or Death From Any Cause
Description: Disease Progression defined as relative decline in 6-minute walking distance (6MWD) from baseline (defined as >25% from baseline or 15-25% from baseline associated with worsening oxygen saturation, worsening Borg score, or increased oxygen requirements), respiratory-related non-elective hospitalizations, or all-cause mortality.
Time Frame: Baseline up to Week 52
Population: Participants with data available at week 52.
Measure: Number; unit: Percentage of Participants
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 88 | 89
Percentage of Participants | 72.7 | 69.7
Statistical Analysis 1: Comparison: Pirfenidone+Sildenafil vs Pirfenidone+Placebo; Test type: Superiority; p = 0.6527, Chi-squared; Difference of percentage of participants = 3.06, 95% CI 2-sided [-11.30 to 17.97]

2. Secondary Outcome: Time to First Occurrence of Disease Progression
Description: Disease Progression defined as relative decline in 6MWD from baseline (defined as >25% from baseline or 15-25% from baseline associated with worsening oxygen saturation, worsening Borg score, or increased oxygen requirements), respiratory-related non-elective hospitalizations, or all-cause mortality.
Time Frame: Baseline up to Week 52
Population: Participants with data available at week 52.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 88 | 89
Weeks | 26.00 [20.57 to 38.14] | 25.43 [13.00 to 37.71]
Statistical Analysis 1: Comparison: Pirfenidone+Sildenafil vs Pirfenidone+Placebo; Test type: Superiority; p = 0.7568, Log Rank; Log-rank test based on the time to the first event to compare the two treatment arms; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.67 to 1.34]

3. Secondary Outcome: Time to Multiple Occurrence of Disease Progression Events
Description: Disease Progression defined as relative decline in 6MWD from baseline (defined as >25% from baseline or 15-25% from baseline associated with worsening oxygen saturation, worsening Borg score, or increased oxygen requirements), respiratory-related non-elective hospitalizations, or all-cause mortality. In case participant had more than one event as described in the endpoint definition the second, third etc event was counted as well for the calculation of the endpoint.
Time Frame: Baseline up to Week 52
Population: Participants with data available at week 52.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 88 | 89
Weeks | 20.57 [13.14 to 26.43] | 13.29 [12.71 to 23.29]
Statistical Analysis 1: Comparison: Pirfenidone+Sildenafil vs Pirfenidone+Placebo; Test type: Superiority; p = 0.3760, Log Rank; Log-rank test based on the time to the first event to compare the two treatment arms; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.68 to 1.15]

4. Secondary Outcome: Percentage of Participants With Decline From Baseline in 6-minute Walking Distance (6MWD) of >= 15%
Time Frame: Baseline up to Week 52
Population: Participants with data available at week 52 to calculate a change from baseline.
Measure: Number; unit: Percentage
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 88 | 89
Percentage | 53.4 | 50.6
Statistical Analysis 1: Comparison: Pirfenidone+Sildenafil vs Pirfenidone+Placebo; Test type: Superiority; p = 0.7046, Chi-squared; Difference (95% CI) = 2.85, 95% CI 2-sided [-12.13 to 17.84]

5. Secondary Outcome: Time to First Occurrence of Relevant ≥15% Decline From Baseline in 6-minute Walking Distance (6MWD)
Time Frame: Baseline up to Week 52
Population: Participants with data available at week 52 to calculate a change from baseline.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 88 | 89
Weeks | 39.00 [27.86 to 52.14] | 38.71 [25.14 to 52.57]
Statistical Analysis 1: Comparison: Pirfenidone+Sildenafil vs Pirfenidone+Placebo; Test type: Superiority; p = 0.7550, Log Rank; Difference (95% CI) = 0.94, 95% CI 2-sided [0.62 to 1.41]

6. Secondary Outcome: Time to Respiratory-Related Non-Elective Hospitalization From Baseline to Week 52
Description: N.A. = non-calculable
Time Frame: Baseline up to Week 52
Population: Participants with data available at week 52.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 88 | 89
Weeks | 54.29 [36.29 to NA] — Insufficient number of participants with events. | NA [42.14 to NA] — Insufficient number of participants with events.
Statistical Analysis 1: Comparison: Pirfenidone+Sildenafil vs Pirfenidone+Placebo; Test type: Superiority; p = 0.9174, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.65 to 1.61]

7. Secondary Outcome: Time to All-Cause Non-Elective Hospitalization
Description: N.A. = non-calculable
Time Frame: Baseline up to Week 52
Population: Participants with data available at week 52.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 88 | 89
Weeks | 47.57 [28.00 to NA] — Insufficient number of participants with events | 49.86 [32.00 to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: Pirfenidone+Sildenafil vs Pirfenidone+Placebo; Test type: Superiority; p = 0.7748, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.70 to 1.62]

8. Secondary Outcome: Time to Death From Any Cause
Time Frame: Baseline up to Week 52
Population: Participants with data available at week 52.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 88 | 89
Weeks | NA [54.43 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: Pirfenidone+Sildenafil vs Pirfenidone+Placebo; Test type: Superiority; p = 0.4258, Log Rank; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.38 to 1.50]

9. Secondary Outcome: Percentage of Participants With Lung Transplantation
Time Frame: Baseline up to Week 52
Population: Participants with data available at week 52.
Measure: Number; unit: Percentage
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 88 | 89
Percentage | 10.2 | 6.7

10. Secondary Outcome: Time to Respiratory-Related Death
Time Frame: Baseline up to Week 52
Population: Participants with data available at week 52.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 88 | 89
Weeks | NA [54.43 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: Pirfenidone+Sildenafil vs Pirfenidone+Placebo; Test type: Superiority; p = 0.3161, Log Rank; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.31 to 1.47]

11. Secondary Outcome: Change From Baseline to Week 52 in Transthoracic Echocardiography (ECHO) Parameter: Peak Tricuspid Regurgitation Velocity
Time Frame: Baseline, Week 52
Population: Participants with data available at week 52 to calculate a change from baseline.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 38 | 29
m/s | -0.014 (0.6326) | 0.103 (0.6699)

12. Secondary Outcome: Change From Baseline to Week 52 in Transthoracic Echocardiography (ECHO) Parameter: Pulmonary Artery Pressure (PAPs)
Time Frame: Baseline, Week 52
Population: Participants with data available at week 52 to calculate a change from baseline.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 41 | 30
mmHg | 2.0 (15.65) | 3.6 (22.38)

13. Secondary Outcome: Change From Baseline to Week 52 in Transthoracic Echocardiography (ECHO) Parameter: Tricuspid Annular Plane Systolic Excursion (TAPSE)
Time Frame: Baseline, Week 52
Population: Participants with data available at week 52 to calculate a change from baseline.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 30 | 27
cm | -0.204 (0.4170) | -0.146 (0.4453)

14. Secondary Outcome: Change From Baseline to Week 52 in Transthoracic Echocardiography (ECHO) Parameter: Right Ventricle Basal Diameter
Time Frame: Baseline, Week 52
Population: Participants with data available at week 52 to calculate a change from baseline.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 29 | 24
cm | 0.462 (1.2305) | 0.095 (1.2875)

15. Secondary Outcome: Change From Baseline to Week 52 in Transthoracic Echocardiography (ECHO) Parameter: Inferior Vena Cava Diameter
Time Frame: Baseline, Week 52
Population: Participants with data available at week 52 to calculate a change from baseline.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 24 | 22
cm | -0.05 (0.595) | -0.09 (0.540)

16. Secondary Outcome: Change From Baseline to Week 52 in Transthoracic Echocardiography (ECHO) Parameter: Left Ventricular Ejection Fraction (LVEF)
Time Frame: Baseline, Week 52
Population: Participants with data available at week 52 to calculate a change from baseline.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 43 | 30
Percentage | 1.22 (9.166) | -0.85 (5.767)

17. Secondary Outcome: Change From Baseline to Week 52 in Carbon Monoxide Diffusing Capacity/ Pulmonary Diffusing Capacity (DLCO)
Time Frame: Baseline, Week 52
Population: Participants with data available at week 52 to calculate a change from baseline.
Measure: Mean (Standard Deviation); unit: Percentage Predicted
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 43 | 29
Percentage Predicted | -2.918 (6.2296) | -2.440 (8.2820)

18. Secondary Outcome: Change From Baseline to Week 52 in Forced Vital Capacity (FVC)
Time Frame: Baseline, Week 52
Population: Participants with data available at week 52 to calculate a change from baseline.
Measure: Mean (Standard Deviation); unit: Percentage Predicted
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 45 | 33
Percentage Predicted | -2.761 (7.8044) | -1.616 (11.1158)

19. Secondary Outcome: Percentage of Participants by World Health Organization (WHO) Functional Class at Week 52
Description: The World Health Organisation (WHO) functional class system defines the severity of an participant's symptoms.
  Class II - Participants with Pulmonary Hypertension resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity causes undue breathlessness, fatigue (tiredness), or activities that can cause chest pain, dizziness or even black outs.
  Class III - Participants with Pulmonary Hypertension resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes undue breathlessness, fatigue (tiredness), or activities that can cause chest pain, dizziness or even black outs.
  Class IV - participants with pulmonary hypertension with inability to carry out any physical activity without symptoms. These participants manifest signs of right heart failure, breathlessness and /or fatigue, which may even be present at rest. Discomfort is increased by any physical activity.
Time Frame: Week 52
Population: Participants with data available at week 52.
Measure: Number; unit: Percentage
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 49 | 36
Percentage
  Class II | 19.3 | 13.5
  Class III | 33.0 | 24.7
  Class IV | 3.4 | 1.1
  Missing | 0 | 1.1

20. Secondary Outcome: Change From Baseline in N-terminal Pro-Brain Natriuretic Peptide (NT-proBNP) Level (pg/mL) at Week 52
Time Frame: Baseline, Week 52
Population: Participants with data available at week 52 to calculate a change from baseline.
Measure: Mean (Standard Deviation); unit: pg/mL)
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 44 | 28
pg/mL) | 110.1 (612.98) | 605.9 (1273.19)
Statistical Analysis 1: Comparison: Pirfenidone+Sildenafil vs Pirfenidone+Placebo; Test type: Superiority; p = 0.5646, Linear Mixed Effects Model; Difference in mean change from baseline = -206.59, 95% CI 2-sided [-920.03 to 506.85]

21. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ) Changes From Baseline at Week 52
Description: The SGRQ is a 50-item questionnaire developed to measure health status (quality of life) in participants with diseases of airways obstruction. Three component scores are calculated, where the higher the component result the worse the condition:
  Symptoms concerned with the effect of respiratory symptoms, their frequency and severity (range: 0-16.61) Activity concerned with activities that cause or are limited by breathlessness (range: 0-30.31) Impacts covers a range of aspects concerned with social functioning and psychological disturbances resulting from airway disease (range: 0- 53.08) Total score summaries the impact of disease on overall health status. Scores are expressed as a percentage of overall impairment where 100 represents worst possible health status and 0 indicates best possible health status.
Time Frame: Baseline, Week 52
Population: Participants with data available at week 52 to calculate a change from baseline.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 41 | 31
Units on a scale
  Total score: number analyzed (Participants) | 41 | 30
  Total score | 6.149 (12.3407) | 11.437 (12.5187)
  Symptoms component score: number analyzed (Participants) | 41 | 30
  Symptoms component score | 2.498 (19.6074) | 8.261 (19.5558)
  Activities component score: number analyzed (Participants) | 41 | 30
  Activities component score | 3.997 (15.4341) | 10.871 (14.5246)
  Impacts component score | 8.417 (15.0040) | 12.118 (15.3487)
Statistical Analysis 1: Comparison: Pirfenidone+Sildenafil vs Pirfenidone+Placebo; Test type: Superiority; p = 0.5255, ANCOVA; Difference in mean change in total score: -4.22; Median Difference (Final Values) = -3.33, 95% CI 2-sided [-9.98 to 2.36]

22. Secondary Outcome: University of California, San Diego-Shortness of Breath Questionnaire (UCSD-SOBQ) Changes From Baseline at Week 52
Description: The UCSD-SOBQ is a respiratory questionnaire and it assesses dyspnea associated with activities of daily living (ADL). Participants indicate severity of SOB on a 6-point scale in 21 ADL. Three additional questions ask about fear of harm from overexertion, limitations and fear caused by SOB. A total score ranges from 0 to 120, with higher scores indicating greater impairment.
Time Frame: Baseline, Week 52
Population: Participants with data available at week 52 to calculate a change from baseline.
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 35 | 25
Points on scale | 12.5 (20.93) | 18.8 (19.68)
Statistical Analysis 1: Comparison: Pirfenidone+Sildenafil vs Pirfenidone+Placebo; Test type: Superiority; p = 0.4263, ANCOVA; Difference in mean change in total score: -5.07; Median Difference (Final Values) = -6.00, 95% CI 2-sided [-18.00 to 6.00]

23. Secondary Outcome: Change From Baseline in Distance Walked, 6-minute Walking Distance (6MWD) Test at Week 52
Time Frame: Baseline up to Week 52
Population: Participants with data available at week 52 to calculate a change from baseline.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 42 | 30
meters | -52.9 (121.07) | -40.8 (91.26)

24. Secondary Outcome: Change From Baseline in Oxygen Requirements, 6-minute Walking Distance (6MWD) Test at Week 52
Time Frame: Baseline up to Week 52
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 42 | 30
L | 0.6 (1.27) | 0.6 (1.43)

25. Secondary Outcome: Change From Baseline in Other 6-minute Walking Distance (6MWD) Parameters at Week 52
Time Frame: Baseline up to Week 52
Population: Participants with data available at week 52 to calculate a change from baseline.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 42 | 30
Percentage
  SpO2 before the test (at rest) | -0.5 (4.63) | -0.8 (3.77)
  SpO2 lowest during the test: number analyzed (Participants) | 20 | 15
  SpO2 lowest during the test | -3.4 (8.93) | 0.3 (5.27)
  SpO2 after the test | 0.5 (9.97) | -2.3 (6.67)

26. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: Baseline up to Week 52 + 28 days
Population: Participants with AEs that started or worsened on or after first intake of randomized treatment until last positive dose + 28 days
Measure: Number; unit: Percentage
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 88 | 89
Percentage | 98.9 | 93.3

27. Secondary Outcome: Borg Scale Result at the End of the Test at Week 52
Description: The Borg Scale rates participant's level of perceived exertion during any activity from 0-10, with 0 being no effort at all and 10 being maximal exertion.
Time Frame: Week 52
Population: Participants with data available at week 52.
Measure: Mean (Standard Deviation); unit: Points on Scale
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
Number analyzed (Participants) | 42 | 30
Points on Scale | 0.9 (3.00) | 0.7 (3.24)

ADVERSE EVENTS:
Time Frame: From baseline to primary data cut-off (up to 2 years 7 months). The safety data includes DBP and SFU up to 11-Nov-2019.
Description: Total # of Deaths (all causes n= 64) represent deaths occurring during Double blind treatment period+4 week FU+additional safety follow up to the database snapshot of 11-Nov-2019.
Arm/Group | Pirfenidone+Sildenafil | Pirfenidone+Placebo
All-Cause Mortality (participants affected / at risk) | 28/88 | 36/89
Serious Adverse Events (participants affected / at risk) | 54/88 | 55/89
Other Adverse Events (participants affected / at risk) | 53/88 | 58/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pirfenidone+Sildenafil (N=88) | Pirfenidone+Placebo (N=89)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 5 (5)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 19 (23) | 21 (31)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 4 (4)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 3 (4) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Blindness transient (Eye disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster disseminated (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1)
Pneumonia (Infections and infestations) | 7 (9) | 4 (4)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (3)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (5)
Lung transplant (Surgical and medical procedures) | 1 (1) | 1 (1)
Cryoglobulinaemia (Vascular disorders) | 0 (0) | 1 (1)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pirfenidone+Sildenafil (N=88) | Pirfenidone+Placebo (N=89)
Diarrhoea (Gastrointestinal disorders) | 11 (15) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5) | 3 (3)
Fatigue (General disorders) | 8 (8) | 6 (6)
Oedema peripheral (General disorders) | 3 (4) | 5 (5)
Bronchitis (Infections and infestations) | 6 (6) | 9 (15)
Influenza (Infections and infestations) | 2 (2) | 5 (6)
Respiratory tract infection (Infections and infestations) | 9 (11) | 4 (6)
Upper respiratory tract infection (Infections and infestations) | 8 (9) | 2 (4)
Weight decreased (Investigations) | 5 (5) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 9 (9)
Dizziness (Nervous system disorders) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 6 (7) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 9 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 (23) | 17 (18)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (6)
Hypotension (Vascular disorders) | 6 (7) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT02951429/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT02951429/SAP_001.pdf